CLINICAL TRIAL: NCT04918667
Title: A Phase I, Randomized, Crossover, Double-blind, Pharmacokinetic Study of Berberine Released From Cyclodextrin in Healthy Volunteers
Brief Title: Effect of Gamma-cyclodextrin on the Bioavailability of Berberine
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EuroPharma, Inc. (Industry)
Collaborators: Scientific Center of Drug and Medical Technologies Expertise of the Ministry of Health, Armenia (Unknown); Cardiomed LLC, Armenia (Unknown); Institute of Fine Organic Chemistry of the National Academy of Science, Armenia (Unknown); Phytomed AB, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP-1007
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Drug Absorption
Keywords: Berberine; gamma-cyclodextrin; Pharmacokinetic; Bioavailability; Berberine MetX™ Ultra Absorption
MeSH Terms: interventions — gamma-cyclodextrin; Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine MetX™ Ultra Absorption (Experimental): 16 healthy subjects will receive orally 500 mg of berberine in two capsules of Berberine MetX™ Ultra Absorption.
  Interventions: Combination Product: Berberine incorporated in gamma cyclodextrin
- Berberine MetX™ (Active Comparator): 16 healthy subjects will receive orally 500 mg of berberine in one capsule of Berberine MetX™ (reference product).
  Interventions: Dietary Supplement: Berberine

INTERVENTIONS:
Combination Product: Berberine incorporated in gamma cyclodextrin — Experimental modified product. One capsule contains 250 mg of Berberine from Indian Barberry (Berberis aristate DC.) Bark and Root Extract incorporated in gamma-cyclodextrin
  Other Names: Berberine MetX™ Ultra Absorption, 250 mg
  Arms: Berberine MetX™ Ultra Absorption
Dietary Supplement: Berberine — Active comparator. One capsule contains 500 mg of Berberine from Indian Barberry (Berberis aristate DC.) Bark and Root Extract
  Other Names: Berberine MetX™, 500 mg
  Arms: Berberine MetX™

SUMMARY:
In this study, we will evaluate the relative bioavailability of Berberine (BB) from capsules containing Indian Barberry (Berberis aristate DC.) Bark and Root Extract in the blood plasma of healthy subjects after oral administration of:

A. Capsules containing Berberine and GCD (BBA Berberine MetX™ Ultra Absorption, 250 mg) B. Capsules containing Berberine (BB, Berberine MetX™, 500 mg) - (reference product).

DETAILED DESCRIPTION:
Study Background

A growing body of evidence suggests that gamma-cyclodextrin (GCD) can increase the clinical efficacy of water-insoluble biologically active compounds with low bioavailability. GCD is the most bio adaptable and helpful to increase the absorption of many drugs, including Berberine from Indian Barberry (Berberis aristate DC.) Bark and Root Extract by forming inclusion complexes or GCD/drug conjugates.

Berberine has been recommended in traditional practice and recognized by modern science to support healthy blood sugar†, cholesterol and triglyceride levels, and overall metabolic health. But despite these findings, standard Berberine can still be difficult for the body to absorb and use effectively.

It's estimated that only about five percent of any given dosage of Berberine makes it into the bloodstream, so finding a way to enhance absorption is key to the full advantage of its benefits.

Hypothesis: gamma-cyclodextrin increases absorption and bioavailability of Berberine from Berberine MetX™ Ultra Absorption capsules.

The study aims to provide experimental evidence supporting or rejecting this hypothesis.

This will be a double-blind, crossover design, pharmacokinetic study, where 16 healthy human volunteers will be randomly assigned to receive two different formulations BBA, and BB, in two consecutive phases of the study:

* Phase A. All patients take capsules BBA., provide blood samples in 0.5, 0.75, 1, 2, 4, 6, 12, 24, and 48 hours (9 points) after administration following washout period for two weeks.
* Phase B. All patients take capsules BB, provide blood samples in 0.5, 0.75, 1, 2, 4, 6, 12, 24, and 48 hours (9 points) after administration following washout period for two weeks.

Subjects will be in the clinic from not less than 11 hours pre-dose to ensure at least 10 hours fasting before administering the investigational product. They will remain in the facility post-dose until at least 24 hours each period, provided they are not suffering from any adverse event.

The concentration of Berberine in all blood samples will be determined using a validated for a limit of detection, accuracy, and precision analytical method (HPLC-MS) with the internal standard - digoxin. Appropriate mathematical methods and Kinetic 4.4.1 software will be used to generate basic pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, as determined by medical history, physical examination, and clinical laboratory testing,
* Willingness to stay in the unit overnight for the duration of the study,
* Provide a signed written informed consent.

Exclusion Criteria:

* overweight (BMI >35 kg/m2),
* pregnancy,
* lactation,
* drug abuse,
* use of dietary supplements or any form of medication (with the exception of oral contraceptives),
* heavy smokers, or ex-smokers with a remote history (> one pack/day),
* frequent alcohol consumption (>20 g ethanol/d),
* adherence to a restrictive dietary regimen,
* physical activity of more than 5 h/wk,
* respiratory tract infections, or suspicion thereof in the last 14 days before dosing,
* history or presence of disease in the kidneys and heart, lungs, liver, gastrointestinal tract, endocrine organs or other conditions such as metabolic disease known to interfere with the absorption, distribution, metabolism, and excretion of drugs,
* malignancy,
* autoimmune disorders such as (but not limited to) lupus erythematosus, multiple sclerosis, rheumatoid arthritis, or sarcoidosis,
* any other disease or condition, which, in the opinion of the Investigator, would make the subject unsuitable for this study,
* currently taking medications known to be CYP2C9 inducers (i.e., carbamazepine and rifampicin).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The area under the plasma concentration versus time curve (AUC, expressed in ng x h/mL) of berberine incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72 and 96 hours, post-dose
  The changes from the baseline the concentration (ng/ml) of berberine in blood plasma obtained after oral administration of the experimental product BBA.
The area under the plasma concentration versus time curve (AUC, expressed in ng x h/mL) of berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72 and 96 hours, post-dose
  The changes from the baseline the concentration (ng/ml) of berberine in blood plasma obtained after oral administration of the active comparator BB.

SECONDARY OUTCOMES:
The absorption rate constants (Ka, h-1) of berberine incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72 and 96 hours, post-dose
  The absorption rate constants (Ka, h-1) of berberine obtained after oral administration of the experimental modified product BBA.
The absorption rate constants (Ka, h-1) of berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72 and 96 hours, post-dose
  The absorption rate constants (Ka, h-1) of berberine obtained after oral administration of the active comparator BB.
Maximum plasma concentration (Cmax, ng/ml) of Berberine incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  Maximum plasma concentration (Cmax, ng/ml), of berberine obtained after oral administration of the experimental modified product BBA
Maximum plasma concentration (Cmax, ng/ml) of Berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  Maximum plasma concentration (Cmax, ng/ml), of berberine - obtained after oral administration of the active comparator BB.
Time to reach maximum plasma concentration, Tmax (h) of berberine incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  Time to reach maximum plasma concentration, Tmax (h) of berberine obtained after oral administration of the experimental modified product BBA
Time to reach maximum plasma concentration, Tmax (h) of berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  Time to reach maximum plasma concentration, Tmax (h) of berberine obtained after oral administration of the active comparator BB.
Mean absorption time MAT (h) of berberine incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  Mean absorption time MAT (h) of berberine obtained after oral administration of the experimental modified product BBA
Mean absorption time MAT (h) of berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  Mean absorption time MAT (h) of berberine obtained after oral administration of the active comparator BB

OTHER OUTCOMES:
Relative bioavailability (%) of berberine incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  Relative bioavailability (%) of Berberine from 0 to 96 hours defined as the ratio of AUC0-96h for the tested formulation (Berberine MetX™ Ultra Absorption capsules) to the AUC0-96h obtained for the reference product (100%, Berberine MetX™ Ultra capsules), given by the same route of administration in the same dose. F= AUCBBA/AUCBB x 100%
Effect of gamma-cyclodextrin on absorption rate constant (Ka, h-1) of berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  The difference in the absorption rate constants (Ka, h-1) of berberine obtained after oral administration of BBA, and BB.
Effect of gamma-cyclodextrin on the maximal concentration (ng/ml) of berberine in blood | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  The difference in Cmax (ng/ml) of berberine obtained after oral administration of BBA and BB.
Effect of gamma-cyclodextrin on time (h) to reach maximum plasma concentration of berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  The difference in Tmax (h) of berberine obtained after oral administration of BBA, and BB.
Effect of gamma-cyclodextrin on Mean absorption time (h) of berberine | 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72, and 96 hours, post-dose
  The difference in MAT (h) of berberine obtained after oral administration of BBA, and BB.

CONTACTS AND LOCATIONS:
Overall Officials: Aghavni Ginosyan, PhD, MD, Principal Investigator — Scientific Center of Drug and Medical Technologies Expertise of the Ministry of Health, Armenia; Samvel Hairumyan, PhD, MD, Principal Investigator — CARDIOMED Family Health Center, LLC of the Ministry of Health of the Republic of Armenia; Areg Hovhannisyan, PhD, Principal Investigator — Institute of Fine Organic Chemistry of the National Academy of Science, Armenia; Alexander G Panossian, PhD, Study Director — Phytomed AB, Sweden
Locations (4):
- Armenia (3):
  - CARDIOMED Family Health Center, LLC of the Ministry of Health of the Republic of Armenia, Yerevan
  - Institute of Fine Organic Chemistry of the National Academy of Science, Yerevan
  - Scientific Center of Drug and Medical Technologies Expertise, Yerevan
- Phytomed AB, Våxtorp, HL, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu CS, Zheng YR, Zhang YF, Long XY. Research progress on berberine with a special focus on its oral bioavailability. Fitoterapia. 2016 Mar;109:274-82. doi: 10.1016/j.fitote.2016.02.001. Epub 2016 Feb 2. PMID 26851175
- [Background] Xu X, Yi H, Wu J, Kuang T, Zhang J, Li Q, Du H, Xu T, Jiang G, Fan G. Therapeutic effect of berberine on metabolic diseases: Both pharmacological data and clinical evidence. Biomed Pharmacother. 2021 Jan;133:110984. doi: 10.1016/j.biopha.2020.110984. Epub 2020 Nov 10. PMID 33186794
- [Background] Loftsson T, Moya-Ortega MD, Alvarez-Lorenzo C, Concheiro A. Pharmacokinetics of cyclodextrins and drugs after oral and parenteral administration of drug/cyclodextrin complexes. J Pharm Pharmacol. 2016 May;68(5):544-55. doi: 10.1111/jphp.12427. Epub 2015 Jun 9. PMID 26059798
- [Background] Kamigauchi M, Kawanishi K, Ohishi H, Ishida T. Inclusion effect and structural basis of cyclodextrins for increased extraction of medicinal alkaloids from natural medicines. Chem Pharm Bull (Tokyo). 2007 May;55(5):729-33. doi: 10.1248/cpb.55.729. PMID 17473458
- [Background] Hopwood VL, Pathak S. Improved quality of Giemsa banding by the use of trypsin concentrate. Am Biotechnol Lab. 1994 Oct;12(11):52. No abstract available. PMID 7765426
- [Background] Tannous M, Caldera F, Hoti G, Dianzani U, Cavalli R, Trotta F. Drug-Encapsulated Cyclodextrin Nanosponges. Methods Mol Biol. 2021;2207:247-283. doi: 10.1007/978-1-0716-0920-0_19. PMID 33113141
- [Background] Uekama K. Design and evaluation of cyclodextrin-based drug formulation. Chem Pharm Bull (Tokyo). 2004 Aug;52(8):900-15. doi: 10.1248/cpb.52.900. PMID 15304981